CLINICAL TRIAL: NCT01902303
Title: Evaluation of Cold Sore Treatments on UV Induced Cold Sores
Brief Title: Evaluation of Cold Sore Treatments on Ultra Violet (UV) Induced Cold Sores
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beech Tree Labs, Inc. (Industry)
Collaborators: Norwich Clinical Research Associates Ltd. (Other); Hill Top Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BTL - 2013-06-0161; HTR - 13-131178 (Other: Hill Top Research)
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-03

CONDITIONS: Oral Herpes Simplex
Keywords: Herpes Labialis; Herpes Simplex; Herpes; Ultra Violet (UV) Induced
MeSH Terms: conditions — Stomatitis, Herpetic; Herpes Labialis; Herpes Simplex

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Matching Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Matching Placebo
- BTL-TML-HSV (Experimental): Experimental Product
  Interventions: Drug: BTL-TML-HSV

INTERVENTIONS:
Drug: Matching Placebo — Sublingual micro dosing of placebo for 7 days
  Arms: Matching Placebo
Drug: BTL-TML-HSV — Sublingual micro dosing of BTL-TML-HSV for 7 days
  Arms: BTL-TML-HSV

SUMMARY:
The purpose of this study is to determine if a new drug treatment is effective to block the development of a cold sore lesion following Ultra Violet (UV) exposure.

DETAILED DESCRIPTION:
This was a multi-center, randomized, evaluator and subject-blind, placebo controlled study design

The objective of this study was to evaluate the ability of the test articles to block the development of a cold sore lesion from progressing beyond the prodromal stage following a UV-induced process.

The primary efficacy endpoint of this study was to determine if a recurrent oral herpes episode initiated with prodromal symptoms was aborted before progressing to a lesion (vesicle) via assessing lesion stages by a trained evaluator.

The secondary efficacy endpoints included: a) subject self-assessments and b) test article weights and diaries to track treatment compliance.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history of recurrent cold sores averaging 2 or more episodes per year
* UV exposure is known to cause a cold sore outbreak

Exclusion Criteria:

* History of abnormal reactions to sunlight
* Used antiviral therapy directly prior to entering study
* Any other condition which in the opinion of the Investigator may affect the results or place the subject at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McMichael, PhD, Study Director — President, Beech Tree Labs, Inc.
Locations (3):
- United States (3):
  - Hill Top Research, St. Petersburg, Florida
  - Hill Top Research, Cincinnati, Ohio
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mamber SW, Hatch T, Miller CS, Murray JV, Strout C, McMichael J. Low-dose Oral Thimerosal for the Treatment of Oral Herpes: Clinical Trial Results and Improved Outcome After Post-hoc Analysis. J Evid Based Integr Med. 2022 Jan-Dec;27:2515690X221078004. doi: 10.1177/2515690X221078004. PMID 35142535

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from 29Jul2013 through 09Sep2014. Subjects were recruited through three research clinics located in the US who had been trained in UVr application used to trigger recurrent oral Herpes Simplex Labialis.
Pre-assignment Details: Subjects who did not meet inclusion/exclusion or withdrew consent prior to enrollment were not enrolled in the study. Eligible subjects underwent minimum erythema dose (MED) UVr determination and if MED criteria was met were randomized. Those enrolled who did not develop prodrome following the UVr induced process were not treated.
Groups:
- Matching Placebo: Matching Placebo
  Treatment regimens will be as follows (upon the first signs/symptoms of prodrome (tingling, itching, burning):
  * Day 0 - Take 1 drop every 10 minutes for the 1st hour following appearance of prodrome symptoms (0, 10, 20, 30, 40, 50 and 60 minutes), then 1 drop every hour until bedtime.
  * Days 1 & 2 - Take 1 drop six times daily -
  * Days 3-7 - Take one drop twice daily
- BTL-TML-HSV: Experimental Product
  BTL-TML-HSV: Sublingual micro dosing of BTL-TML-HSV for 7 days
  Treatment regimens will be as follows (upon the first signs/symptoms of prodrome (tingling, itching, burning):
  * Day 0 - Take 1 drop every 10 minutes for the 1st hour following appearance of prodrome symptoms (0, 10, 20, 30, 40, 50 and 60 minutes), then 1 drop every hour until bedtime.
  * Days 1 & 2 - Take 1 drop six times daily -
  * Days 3-7 - Take one drop twice daily
Period: Overall Study
Arm/Group | Matching Placebo | BTL-TML-HSV
Started | 77 (Allocated to placebo) | 81 (Allocated to active treatment)
Number of Participants | 56 (Number of randomized participants who developed a cold sore and used the assigned treatment.) | 62 (Number of randomized participants who developed a cold sore and used the assigned treatment.)
Completed | 54 (21 not treated - did not use placebo medication as they did not develop cold sore) | 57 (19 not treated /did not use medication as they did not develop a cold sore)
Not Completed | 23 | 24
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 2 | 2
Not completed — subject lost investigational product | 0 | 1
Not completed — Did not develop a cold sore | 21 | 19

BASELINE CHARACTERISTICS:
Population: Demographics based on number of subjects who were randomization and subsequently assigned investigational product
Groups:
- Matching Placebo: Placebo Safety Population - All subjects enrolled and received placebo test article
- BTL-TML-HSV Active Treatment: BTL-TML Safety Population - All subjects enrolled and received active test article
- Total: Total of all reporting groups
Arm/Group | Matching Placebo | BTL-TML-HSV Active Treatment | Total
Number analyzed (Participants) | 77 | 81 | 158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 72 | 73 | 145
  >=65 years | 5 | 8 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 57 | 115
  Male | 19 | 24 | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants for Whom a Recurrent Oral Herpes Episode Initiated With Prodromal Symptoms Were Aborted Before Progressing to a Lesion as Assessed by a Trained Evaluator
Description: The primary efficacy endpoint of this study is to determine if a recurrent oral herpes episode initiated with prodromal symptoms is aborted before progressing to a lesion (vesicle stage) via assessing lesion stages by the trained evaluator. Any episode of oral herpes that did not reach a vesicle stage or higher by Day 7 (based on evaluator and self-assessments of legion stage) was considered "aborted" or "blocked". Any episode of oral herpes that reached a vesicle stage or higher by Day 7 was considered a treatment failure.
Time Frame: Day 0- Day 7
Population: Participants that did not experience prodrome stage as assessed by the evaluator or met major protocol violations were not included in the PP analysis.
Measure: Number; unit: participants who had aborted lesions
Groups:
- Matching Placebo: Placebo Efficacy Population - All subjects enrolled and received placebo test article and met Per protocol definition
- BTL-TML-HSV Active Treatment: BTL-TML Efficacy Population - All subjects enrolled and received active test article and met Per Protocol definition
Arm/Group | Matching Placebo | BTL-TML-HSV Active Treatment
Number analyzed (Participants) | 14 | 23
participants who had aborted lesions | 6 | 11
Statistical Analysis 1: Comparison: Matching Placebo vs BTL-TML-HSV Active Treatment; Test type: Superiority or Other; p > .5000, Chi-squared

2. Secondary Outcome: Number of Participants for Whom a Recurrent Oral Herpes Episode Initiated With Prodromal Symptoms Were Aborted Before Progressing to a Lesion as Assessed by the Participant
Description: The secondary efficacy endpoint of this study is to determine if a recurrent oral herpes episode initiated with prodromal symptoms is aborted before progressing to a lesion (vesicle stage) via assessing lesion stages by the participant. Any episode of oral herpes that did not reach a vesicle stage or higher by Day 7 (based on evaluator and self-assessments of legion stage) was considered "aborted" or "blocked". Any episode of oral herpes that reached a vesicle stage or higher by Day 7 was considered a treatment failure.
Time Frame: 0 -7 days
Population: 158 subjects randomized to treatment. 118 subjects used allocated assigned treatment (62 test article and 56 placebo). 7 subjects failed to complete and 111 completed study. For this secondary analysis (self assessments) 53 subjects noted prodrome occurring on Day 0.
Measure: Number; unit: participants with aborted lesions
Groups:
- Matching Placebo: Placebo efficacy Population - All subjects who received placebo test article and were compliant with protocol
- BTL-TML-HSV Active Treatment: BTL-TML Efficacy Population - All subjects who received active test article and were compliant with protocol
Arm/Group | Matching Placebo | BTL-TML-HSV Active Treatment
Number analyzed (Participants) | 28 | 25
participants with aborted lesions | 6 | 8
Statistical Analysis 1: Comparison: Matching Placebo vs BTL-TML-HSV Active Treatment; Test type: Superiority or Other; p = .3835, Chi-squared

ADVERSE EVENTS:
Time Frame: AEs were collected from the time of informed consent until end of follow up period which was up to 14 days after start of treatment.
Description: Serious AE were collected for all patients. AEs noted over 5% were only for those patients that took study medication.
Groups:
- Matching Placebo: Placebo Safety Population - All subjects that enrolled and were allocated to placebo test article except for SAEs and that includes all subjects that signed informed consent.
- BTL-TML-HSV Active Treatment: BTL-TML Safety Population - All subjects enrolled and allocated to active test article except for SAEs which includes all subjects that signed informed consent.
Arm/Group | Matching Placebo | BTL-TML-HSV Active Treatment
Serious Adverse Events (participants affected / at risk) | 0/222 | 0/81
Other Adverse Events (participants affected / at risk) | 7/56 | 6/62
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Matching Placebo (N=56) | BTL-TML-HSV Active Treatment (N=62)
Blood pressure diastolic increased (Investigations) | 3 (3) | 4 (4)
Heart rate increased (Investigations) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days